CLINICAL TRIAL: NCT04326218
Title: Immunopathological Analysis in a French National Cohort of Membranous Nephropathy (IHMN)
Brief Title: Immunopathological Analysis in a French National Cohort of Membranous Nephropathy
Acronym: IHMN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 18-GIRCI-03
Record Dates: First submitted 2019-12-26; First posted 2020-03-30 (Actual); Last update posted 2020-04-07 (Actual); Status verified 2020-03

CONDITIONS: Membranous Nephropathy
MeSH Terms: conditions — Glomerulonephritis, Membranous | interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: Descriptive analysis of patient cohort who will be subjected to specific samples related to the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cohort (Other): All patients included will have to be taken blood samples
  Interventions: Other: Blood sample

INTERVENTIONS:
Other: Blood sample — Serum samples will be sent for centralised analyses in Nice.
  On these samples, different analysis will be performed :
  * anti-PLA2R1 and anti-THSD7A antibodies
  * anti-PLA2R1 and anti-THSD7A epitopes
  * HLA typing

SUMMARY:
National cohort of all cases of membranous nephropathy (MN) during a 1 year period in France, based on a pathological and/or serological diagnostic, collecting the data on:

* incidence of MN
* prevalence of anti-PLA2R1 and anti-THSD7A
* clinical outcome one year after diagnosis or after relapse (complete remission, partial remission or persistent nephrotic syndrome)
* environmental risk factors for the onset of MN
* HLA markers
* patient care status in France

DETAILED DESCRIPTION:
Membranous nephropathy is a rare auto-immune disease, yet a major cause of nephrotic syndrome in adults. It is characterised by the deposition of antigen-antibody complexes on the glomerular basement membrane, leading to a decreased filtration rate and eventually kidney failure. About one third of cases have a favourable outcome without any treatment, another third requires a long term symptomatic treatment to manage their symptoms, and the last third of patients advances to end stage renal failure, requiring dialysis and kidney graft. MN can be associated with cancer, infections, other auto-immune diseases and with certain drugs (secondary MN), but most often it is idiopathic. In the latter form two antigens have been identified, PLA2R1 and THSD7A, with corresponding auto-antibodies in 70% and 2% of MN patients, respectively. GWAS studies identified several alleles associated with a higher risk of developing MN, however, since these are common variants they cannot explain the onset of MN in the vast majority of cases. Since MN is a rare disease, the number of new cases per each center is low, and nation-wide studies are needed to correctly evaluate its incidence and risk factors for the onset of MN, as well as validate previously published findings in monocentric studies on the prognostic value of PLA2R1 epitope spreading (immunisation against multiple domains of PLA2R1).

This study aims to establish a French national cohort of all cases of MN in a one year period in France. The inclusion will last one year with one additional year of follow-up, for a total of 2 years. In the first year, nephrologists of each associate centers in France will propose the study to each of their patients diagnosed with MN. In addition, clinical information will be collected, as well as a survey on patients' lifestyle habits. Serum samples will be sent for centralised analyses in Nice.

This study will help to clarify the results from single center studies, such as the prognostic value of epitope spreading. The information acquired on environmental risk factors will help us understand the pathophysiological mechanisms leading to the onset of MN et, by association, to other auto-immune diseases. With this knowledge, measures could be put in place to protect the population at risk.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or more
* Biopsy on a native kidney consistent with MN and/or positivity for serum anti-PLA2R1 and/or anti-THSD7A antibodies
* Signed informed consent

Exclusion Criteria:

* Diagnosis error based on the kidney biopsy staining or on serology analyses for the positivity for anti-PLA2R1 and/or anti-THSD7A
* Patients unable to give an informed consent
* Patients withdrawing an informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2020-07-01 (Estimated); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
To determine the incidence of Membranous Nephropathy (MN) and its evolution | one year after inclusion
  as either complete remission (UPCR < 0.3 g/g, serum albumin > 35 g/L, eGFR > 60 ml/min/1.73 m²) or partial remission (UPCR < 3.5 g/g and reduction of at least 50% from baseline, < 20% increase of serum creatinin from baseline) or persistent nephrotic syndrome (UPCR > 3.5 g/g, serum albumin < 30 g/L)

SECONDARY OUTCOMES:
Determination of incidence of primary and secondary forms of MN | 24 months
Identification of environmental factors associated with the onset of MN | 24 months
  Thanks to a specific questionnaire data on medical history, lifestyle, demography and profession will be collected
  * Medical history: prior diagnosis of any autoimmune disease, cancer, infection or other, infection in the month before the diagnosis of MN, thrombosis, drugs taken at the moment of diagnosis, allergies and type of symptomes
  * Emotional state: emotional state at diagnosis, stressful or destabilizing event in the year preceding diagnosis of MN
Description of the standard of care for patients with MN in France | 24 months
  Treatment names and their duration (in weeks) will be collected
the prognostic value of epitope spreading in patients with PLA2R1-associated MN | 24 months
  Epitope spreading status is determined by measuring the positivity to anti-CysR, anti-CTLD1 and CTLD7 antibodies in the serum, by the means of ELISA and expressed as RU/mL. The patients with antibodies targetting CysR only are considered as non-spreaders, while the patients additionnaly targetting either CTLD1 and/or CTLD7 are considered as spreaders. Epitope spreading status (non-spreader or spreader) will be correlated to clinical outcome (complete remission, partial remission or persistent nephrotic syndrome, as defined under primary outcome measures) one year after inclusion.
Characterization of HLA typing of MN patients | 12 months
  Isolation of DNA and genotyping will be performed with the use of standard procedures of Next Generation Sequencing
Prognostic value of tissue staining for glomerular deposit of PLA2R1, THSD7A, as welle as of different IgG subclasses | 12 months
  Positivity for PLA2R1, THSD7A and NELL-1 antigens will be determined using immunostaining with antibodies against PLA2R1, THSD7A and NELL-1, and Positivity for IgG1 IgG2, IgG3 and IgG4 subclasses will be determined using immunostaining with antibodies against IgG1 IgG2, IgG3 and IgG4, respectively, in glomeruli of kidney biopsy at inclusion. The positivity of tissue staining for PLA2R1, THSD7A and NELL-1or Ig subclasses will be correlated to the patient's clinical outcome one year after inclusion (complete remission, partial remission or persistent nephrotic syndrome, as defined under primary outcome measures).

IPD SHARING:
Plan to Share IPD: No
No data will be shared

REFERENCES:
- [Derived] Cremoni M, Agbekodo S, Teisseyre M, Zorzi K, Brglez V, Benzaken S, Esnault V, Planchard JH, Seitz-Polski B. Toxic Occupational Exposures and Membranous Nephropathy. Clin J Am Soc Nephrol. 2022 Nov;17(11):1609-1619. doi: 10.2215/CJN.02930322. Epub 2022 Oct 25. PMID 36283759